CLINICAL TRIAL: NCT06883331
Title: Validity of Computed Guided Technology in Proper Placement of Intermaxillary Fixation Screws in Mandibular Fractures
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 763/2024; Suez Canal University (Other: ethtical committee of suez canal university)
Record Dates: First submitted 2025-03-12; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-04

CONDITIONS: Mandibular Fractures
Keywords: mandible; fracture; fixation; screws
MeSH Terms: conditions — Mandibular Fractures; Fractures, Bone

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IMF screws without surgical guide (Active Comparator): control group: the patients will be treated without surgical guide, conventionally based on surgeon's clinical Experience.
  Interventions: Procedure: intermaxillary fixation using IMF screws
- IMF screws with a surgical guide (Experimental): study group: the patients will be treated using Computer Assisted Surgical Guide to achieve accurate placement of IMF screws.

INTERVENTIONS:
Procedure: intermaxillary fixation using IMF screws — IMF screws will be placed at the junction of the attached and alveolar mucosa, after verifying the root position on the orthopantomogram (OPG) radiograph. One screw in each quadrant was sufficient; all IMF screws will be placed with the patient under local anesthesia or general anesthesia . Cortical perforation with a 1.5-mm drill bit under copious irrigation will be performed or by self-drilling IMF screws and the IMF screws will be tightened on the drilled hole.
  After IMFS placement, intraoperative IMF will be achieved by passing round, stainless steel wires through the screw head to achieve satisfactory occlusion.
  Other Names: IMF
  Arms: IMF screws without surgical guide
Procedure: intermaxillary fixation using IMF screws with surgical guide — The patient's CBCT images in DICOM format will be converted into stereolithographic (STL) images using the segmentation software.
  The converted CBCT STL images will be integrated to obtain the exact tooth morphology Virtual surgical planning (VSP) will be carried out using software to select the exact position of IMF screws placement away from any vital, anatomical or tooth structure.
  these locations will be incorporated into the patients specific IMF surgical guides as access holes to direct the IMF screws drill.
  Guide will be constructed with a thickness of 2-3 mm and printed using Photopolymer Resin® (Form labs) in the CAD/CAM 3- dimensional (3D) printer

SUMMARY:
A randomized clinical study that aims to assess the validity of the use of computer guided technique in the proper placement of IMF screws in mandibular fractures

DETAILED DESCRIPTION:
Fractures of the facial skeleton involving the teeth bearing segments can lead to disruption of the dental occlusion, and difficulties with speech and mastication. The temporary fixation of opposing jaws is called maxillomandibular fixation and is usually secured through placement of IMF screws and wires. The correct placement of IMF screws can be challenging. Such planning may make use of radiographs and computed tomography scans. Knowledge of safe zones in the facial skeleton for screw placement through the use of pre-operative 3-dimensional planning may prevent some of the cited complications. The use of a custom made surgical guide for IMF screw placement has the potential to reduce operation time, optimize screw position, and minimize injury to dental roots and important anatomical structures. Aim: The aim of this study is to Assess the use of computed guided technique in the proper placement of IMF screws in mandibular fractures. Materials and Methods: This clinical study will be conducted on 20 patients who will be equally and randomly distributed into 2 groups: Group A: 10 patients will be treated with 3D guided placement of IMF screw. Group B: 10 patients will be treated with Conventional placement of IMF screws.

To assess the accuracy of IMF screws placement in each group.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffer from recent mandibular fractures that requires fixation
* Dentulous patients
* Medically fit for surgery (ASA I AND ASA II)

Exclusion Criteria:

* Edentulous patients
* Patient with bone pathosis
* patients with primary and mixed dentition
* pathologic mandibular fracture

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-04-27 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
radiographic evaluation | immediately postoperative
  radiographic follow up of the patients immediate postoperatively with CBCT to assess the accuracy of IMF screws placement.
  CBCT will be assessed to detect any injury to the roots of the teeth adjacent to the IMF screws as well as any injury to the adjacent vital structures

SECONDARY OUTCOMES:
clinical evaluation | intra-operative
  clinical evaluation will be done intra-operatively to assess the time consumed in the study group compared to the control group

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Elsholkamy, Professor, Study Director — Suez Canal University; Yasser N Helmy, Prof, Study Director — Specialized Dental Hospital Kobry el Kobba Military Complex, Military Medical Academy; mohamed H Elsherbiny, Dr, Principal Investigator — Specialized Dental Hospital Kobry el Kobba Military Complex, Military Medical Academy
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Joseph Kamal. 2021. Computer Assisted Guided Placement of IMF Screws in Craniomaxillofacial Trauma: An Evolving Technique, Vol. 2(2) 170-173 DOI: 10.1177/27325016211008654 journals.sagepub.com/home/fac